CLINICAL TRIAL: NCT02745873
Title: Lead Detoxifying Effects of Ascorbic Acid Among School Going Adolescents of Karachi- A Cluster Randomized Control Trial
Acronym: LDVC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Pakistan Science Foundation (Other)
Responsible Party: Principal Investigator, Muhammad Ilyas, Mr., Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LDVC
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Elevated Blood Lead Levels
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Ascorbic Acid 250 mg in tablet form was used.
  Interventions: Drug: Ascorbic Acid
- Arm B (Experimental): Ascorbic Acid 500 mg in tablet form was used.
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — Ascorbic Acid (vitamin-c) 500 mg in tablet form was used.
  Other Names: Vitamin C

SUMMARY:
The toxic nature of lead has been recognized ubiquitous for than 2,000 years and today it is a persistent and common environmental contaminant in most parts of the world. Vitamin C is a strong antioxidant and a metabolic co factor playing an important role in many biological processes and biochemical functions (hydroxylation reactions). The research objective is to assess the effect of oral ascorbic acid supplementation 500mg and 250 mg once a day for 4 weeks on Blood Lead level among school going urban adolescents, using a cluster randomized trial study design. Ascorbic Acid (vitamin C) 250 and 500 mg will be administered in two study arms.

ELIGIBILITY:
Inclusion Criteria:

1-school going adolescents, aged 13-18 years.

Exclusion Criteria:

1. Children with history or presence of chronic illness or bleeding disorders, requiring red blood cell transfusion, dialysis
2. Using multivitamins
3. Those who planning to leave study place within 2 months of start of study

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Blood Lead Level | 4 weeks
  Mean Change in blood lead level is the main outcome of the study. It will be recorded as continuous variable and unit of measurement will be μg/dl.
  Blood lead levels will be assessed at baseline before the start of intervention and at the end of the 4 weeks of intervention period in both arms.
  Mean change will be calculated by taking difference between two the points as follow up (4 weeks) Blood lead levels minus baseline Blood Lead level.